CLINICAL TRIAL: NCT07114003
Title: Effects of Virtual Reality Application on Pain, Anxiety, and Patient Satisfaction in Dressing Patients With Pressure Sores: A Randomized Controlled Trial
Brief Title: Effects of Virtual Reality Application on Pain, Anxiety, and Patient Satisfaction in Dressing Patients With Pressure Sores
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: Toros University (Other)
Responsible Party: Principal Investigator, Derya Gezer, Assistant Professor, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Tarsus University
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Pressure Wounds
Keywords: Virtual Reality; Pain; Anxiety; Patient Satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a two-group, repeated-test design, experimental, randomized controlled interventional study aiming to evaluate the effect of VR application.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental Group) (Experimental): In the experimental group, a distraction-inducing intervention will be performed using virtual reality goggles. Unlike traditional methods, the VR goggle method is designed to provide patients with an interactive experience in a visual and auditory environment. The audio and video content of the VR program will be determined by drawing inspiration from proven studies and consulting with healthcare professionals with clinical experience. This method aims to create a stronger distraction effect and achieve greater effectiveness in pain and anxiety management. Pain levels will be measured from all participants before, during, and after the dressing application; a state anxiety inventory will be completed after the dressing application.
  Interventions: Behavioral: virtual reality application
- Routine Care (Control Group) (No Intervention): All participating patients will be interviewed in the clinic to obtain written informed consent. A personal information form and a state-trait anxiety inventory will be completed. All participants will receive standard treatment and nursing practices during wound care. These practices include proper wound cleaning, use of aseptic techniques for infection control, and thorough implementation of dressing procedures. Additionally, routine distraction methods (e.g., listening to music, talking to the patient, reading a book) are recommended and implemented by the nurses in the clinic, depending on the patient's preference.

INTERVENTIONS:
Behavioral: virtual reality application — The Oculus Meta Quest Pro is a virtual reality headset with 256 GB of storage. Its LCD screen offers a resolution of 1800 x 1920 pixels per eye and supports refresh rates from 90 Hz to 120 Hz. It is powered by a Qualcomm Snapdragon XR2+ processor. It features eye tracking and facial tracking, controllers with TruTouch haptics and precision tracking, and built-in 3D spatial audio support. The program, which will be played through the VR headset, is designed to use licensed programs featuring nature scenes (forest, sea, beach, etc.) and relaxing music for 20-30 minutes. The program content will be created by selecting nature sounds and music known to be effective in reducing stress and anxiety. To ensure the program's internal validity, the opinions of healthcare professionals with clinical experience will be obtained to assess whether the program achieves the intended relaxing effect.
  Arms: Virtual reality (Experimental Group)

SUMMARY:
Pressure ulcers are serious and costly wounds that typically develop as a result of impaired blood flow in tissues exposed to prolonged pressure. They are particularly at risk in the elderly, critically ill patients, and individuals with limited mobility. Pain and anxiety during dressing applications for pressure ulcers can negatively impact patient comfort and compliance. There are limited studies in the literature on the use of nonpharmacological methods to reduce pain and anxiety during the dressing process for pressure ulcers. Virtual reality (VR) applications stand out as an effective method for managing pain and anxiety by providing distraction. However, existing studies generally cover all chronic wounds and lack specific research on the use of VR during the dressing process in individuals with pressure ulcers. Therefore, the proposed study aims to examine the effects of VR application during dressing on pain, anxiety, and patient satisfaction in patients with pressure ulcers and aims to make an original contribution to the literature.

DETAILED DESCRIPTION:
A pressure ulcer is a condition that occurs when local tissues in a patient are subjected to prolonged pressure, affecting blood circulation and causing pathological changes . Individuals exposed to prolonged pressure are at high risk of developing pressure ulcers due to local tissue compression, inadequate nutrition, and soft tissue necrosis. Pressure ulcers typically develop as a result of local factors (e.g., pressure, friction, shear, and/or moisture) acting at the level of bony prominences or mechanical pressure from medical devices (cable, cannula, drain, etc.). However, the formation of these wounds is multifactorial, and individual characteristics (age, comorbidities, nutritional status, etc.) also play an important role. With increasing life expectancy, the risk of pressure ulcers increases in older adults, critically ill patients, and those with spinal cord injury or disease. Despite preventive measures, the incidence of pressure ulcers has not decreased for decades. In addition to the risk of pain, infection, and death, the cost of treating pressure ulcers is also quite high. Therefore, developing practices to prevent and treat pressure ulcers is critical. According to the 2023 guidelines of the Wound Healing Society (WHS) and the European Tissue Repair Society (ETRS), pressure ulcers are frequently painful, and this pain is often associated with dressing changes (Level III). Uncontrolled pain can negatively impact patient compliance and quality of life, leading to anxiety. Kim et al.explained the factors affecting pain in pressure wounds with a proposed conceptual framework derived from the biopsychosocial model and emphasized that wound care nurses should implement interventions to reduce pain and anxiety. The duties of wound care nurses, an important part of the multidisciplinary healthcare team in wound care, are not limited to prevention and treatment strategies; they also encompass responsibilities focused on patient-centered, holistic management. The holistic care practices of wound care nurses have been shown to be generally associated with positive outcomes in terms of wound healing, pressure sore incidence, and treatment costs. Furthermore, the importance of considering the main symptoms frequently experienced by patients, such as pain, anxiety, depression, and stress, has been emphasized for a holistic assessment of wound care. In providing effective pain control, the combined application of both pharmacological and non-pharmacological methods with a multimodal approach is strongly emphasized. The almost complete absence of side effects, low cost, and ease of application of non-pharmacological methods used in pain management provide many advantages, such as saving labor and reducing the frequency of analgesic use. Virtual reality (VR) applications are used as a non-pharmacological treatment option to reduce acute and chronic pain and anxiety. More specifically, it is assumed that VR applications alter the negative emotions associated with previous pain experiences and reframe this experience in a positive way by giving the user the experience of being in a new environment. In the clinical setting, VR can also reduce the level of pain-related anxiety by altering the processing of cognitive and emotional affect signals in the central nervous system. By manipulating the environment, it constitutes an effective emotion-focused coping strategy by shifting the focus of attention away from unpleasant stimuli . The literature reports that VR application has positive effects on wound dressing changes and chronic pain. It has been reported that the use of VR during burn dressings positively affects children's physiological parameters and is effective in reducing fear, anxiety, and pain levels.

To our knowledge, no studies have been found in the literature specifically addressing the use of VR, a non-pharmacological method, in the dressing process of pressure ulcers. In this context, the proposed project makes a unique contribution to the literature by focusing solely on the use of VR in patients with pressure ulcers. In light of these considerations, the aim of this study was to evaluate the effects of VR use on pain and anxiety during dressing in patients with pressure ulcers, as well as patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be individuals aged 18 and over (inclusive), who have no hearing/visual impairment, do not have epilepsy, vertigo, or claustrophobia, and who agree to participate in the study.

Exclusion Criteria:

* Patients who exhibit symptoms of cybersickness (dizziness, nausea, etc.) due to the VR application, who require analgesia during the intervention, or who do not feel pain due to neuropathy, and who express their wish to withdraw from the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | Before the Procedure, during the Procedure (10th minute), and baseline, after an average of 20-30 minutes
  In measuring pain, a visual assessment scale (VAS) will be used, where the evaluation is made by making marks on a 100 mm or 10 cm vertical or horizontal line, where there is no pain at one end and the most severe pain at the other end. Pain will be measured using a visual analog scale (VAS), which uses markings on a 100 mm or 10 cm vertical or horizontal line, with no pain at one end and the most severe pain at the other. Pain will be measured before, during, and after dressing application.
Anxiety Assesment | Before the Procedure and baseline, after an average of 20-30 minutes
  State Trait Anxiety Inventary will be used. Before the dressing, the state and trait anxiety inventories will be administered. After the dressing, the state anxiety inventory will be administered again to assess anxiety. This constant value is 50 for state anxiety and 35 for trait anxiety. The resulting value represents the individual's anxiety score. Interpretation of Scores: The total score obtained from both scales ranges from 20 to 80. A higher score indicates a higher level of anxiety, while a lower score indicates a lower level of anxiety.
Patient satisfaction | baseline, after an average of 20-30 minutes
  Patients will be asked about their satisfaction with the application (not satisfied, undecided, satisfied, very satisfied) and the experimental group will be asked whether they would like to use the SG application again.

CONTACTS AND LOCATIONS:
Overall Officials: Derya GEZER, Asisstant Professor, Principal Investigator — Tarsus University; Esma Gökçe, Asisstant Professor, Study Director — Toros University; Dudu Alptekin, Dr, Principal Investigator — Cukurova University
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Results regarding the effects of VR use on pain, anxiety, and patient satisfaction during dressing of patients with pressure ulcers will be shared. However, your personal information will not be shared.
Supporting Information: CSR

REFERENCES:
- [Background] Kilic U, Tural Buyuk E. The Effect of Using Virtual Reality During Burn Dressing on Pain, Anxiety and Fear Felt in Children: A Randomized Controlled Trial. J Burn Care Res. 2024 Aug 6;45(4):949-957. doi: 10.1093/jbcr/irae005. PMID 38224569
- [Background] Gould LJ, Alderden J, Aslam R, Barbul A, Bogie KM, El Masry M, Graves LY, White-Chu EF, Ahmed A, Boanca K, Brash J, Brooks KR, Cockron W, Kennerly SM, Livingston AK, Page J, Stephens C, West V, Yap TL. WHS guidelines for the treatment of pressure ulcers-2023 update. Wound Repair Regen. 2024 Jan-Feb;32(1):6-33. doi: 10.1111/wrr.13130. Epub 2023 Dec 20. PMID 37970711
- [Background] Gefen A, Alves P, Ciprandi G, Coyer F, Milne C, Ousey K, Ohura N, Waters N, Worsley P, Black J, Barakat-Johnson M, Beeckman D, Fletcher J, Kirkland-Kyhn H, Lahmann NA, Moore Z, Payan Y, Schluer AB. An international consensus on device-related pressure ulcers: SECURE prevention. Br J Nurs. 2020 Mar 12;29(5):S36-S38. doi: 10.12968/bjon.2020.29.5.S36. PMID 32167820
- [Background] Fearns N, Heller-Murphy S, Kelly J, Harbour J. Placing the patient at the centre of chronic wound care: A qualitative evidence synthesis. J Tissue Viability. 2017 Nov;26(4):254-259. doi: 10.1016/j.jtv.2017.09.002. Epub 2017 Sep 5. PMID 28893459
- [Background] Edsberg LE, Black JM, Goldberg M, McNichol L, Moore L, Sieggreen M. Revised National Pressure Ulcer Advisory Panel Pressure Injury Staging System: Revised Pressure Injury Staging System. J Wound Ostomy Continence Nurs. 2016 Nov/Dec;43(6):585-597. doi: 10.1097/WON.0000000000000281. PMID 27749790
- [Background] Dowsett C. T.I.M.E. to improve patient outcomes: use of a clinical decision support tool to optimise wound care. Br J Community Nurs. 2019 Mar 1;24(Sup3):S6-S11. doi: 10.12968/bjcn.2019.24.Sup3.S6. PMID 30817187
- [Background] Coleman S, Gorecki C, Nelson EA, Closs SJ, Defloor T, Halfens R, Farrin A, Brown J, Schoonhoven L, Nixon J. Patient risk factors for pressure ulcer development: systematic review. Int J Nurs Stud. 2013 Jul;50(7):974-1003. doi: 10.1016/j.ijnurstu.2012.11.019. Epub 2013 Feb 1. PMID 23375662
- [Background] Chuan A, Zhou JJ, Hou RM, Stevens CJ, Bogdanovych A. Virtual reality for acute and chronic pain management in adult patients: a narrative review. Anaesthesia. 2021 May;76(5):695-704. doi: 10.1111/anae.15202. Epub 2020 Jul 27. PMID 32720308
- [Background] Choi T, Heo S, Choi W, Lee S. A Systematic Review and Meta-Analysis of the Effectiveness of Virtual Reality-Based Rehabilitation Therapy on Reducing the Degree of Pain Experienced by Individuals with Low Back Pain. Int J Environ Res Public Health. 2023 Feb 16;20(4):3502. doi: 10.3390/ijerph20043502. PMID 36834197
- [Background] Boyko TV, Longaker MT, Yang GP. Review of the Current Management of Pressure Ulcers. Adv Wound Care (New Rochelle). 2018 Feb 1;7(2):57-67. doi: 10.1089/wound.2016.0697. PMID 29392094